CLINICAL TRIAL: NCT02231411
Title: Neonatal Resuscitation With Intact Cord
Acronym: NRIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director Neonatal Research Institute, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NRIC; 5R21HD080594 (NIH)
Record Dates: First submitted 2014-08-11; First posted 2014-09-04 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Intraventricular Hemorrhage
Keywords: Delayed Cord Clamping; Pulmonary Ventilation
MeSH Terms: interventions — Umbilical Cord Clamping; Desiccation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ventilation during DCC (V-DCC) (Active Comparator): Measuring the volume of placental transfusion with ventilation (CPAP 5 cm H2O between inflations) in infants born by C/S or VG using, as an initial surrogate marker, Hematocrits at 12 hours of life (HOL)
  Interventions: Procedure: V-DCC
- DCC plus dry and stimulate (Active Comparator): Measuring the volume of placental transfusions with delayed cord clamping alone (DCC) in infants born by C/S or VD using, as an initial surrogate marker, Hematocrits at 12 hours of life (HOL)
  Interventions: Procedure: Delayed cord clamping; Procedure: Dry and and if apneic initially can stimulate by gently rubbing the back for approximately 30 seconds with warm sterile towels

INTERVENTIONS:
Procedure: V-DCC — Ventilation with CPAP 5 cm H2O between inflations and Delayed clamping of the umbilical cord for 60 seconds
  Arms: Ventilation during DCC (V-DCC)
Procedure: Delayed cord clamping — Delayed clamping of the umbilical cord for 60 seconds
  Arms: DCC plus dry and stimulate
Procedure: Dry and and if apneic initially can stimulate by gently rubbing the back for approximately 30 seconds with warm sterile towels
  Arms: DCC plus dry and stimulate

SUMMARY:
The purpose of this study is to examine whether providing ventilation during delayed umbilical cord clamping provides greater placental transfusion and improved hemodynamic transition at birth.

DETAILED DESCRIPTION:
Subjects will receive 1 minute of delayed cord clamping in both arms. One arm will receive routine care, warm dry and stimulate during the 1 minutes transfusion. The second arm will receive routine care PLUS administration of CPAP and if need positive pressure ventilation. The outcome is to determine whether the addition of ventilation provides a larger placental transfusion and a smoother transition at birth.

ELIGIBILITY:
Inclusion Criteria:

* Gestational Age: Women admitted 23+0 to 31+6 weeks (Reason: Highest risk for IVH)

Exclusion Criteria:

* Gestational Age: Parents decline consent (Reason: Can only perform intervention at time of delivery)
* Congenital anomalies of newborn (Reason: Exclude the effect of abnormal hematological function)
* Placental abruption (Reason: Exclude pregnancies at risk for hemorrhage at the time of delivery)
* Twin to twin transfusion (Reason: Exclude possible loss of blood from other twin during delayed cord clamping)
* Placenta Accreta
* Prolonged premature rupture of membranes (> 2 weeks) prior to 23 weeks gestation

Ages: 23 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Peak Hematocrit | within 24 hours

SECONDARY OUTCOMES:
Maximum inspired oxygen (FiO2) (percentage) | over the first 5 minutes of life
Positive Pressure Ventilation given | 1 minute
DR interventions after delayed cord clamping complete | 10 minutes of life
  PPV, CPAP, intubation, chest compressions, volume, medications (yes/no)
Maximum Peak Inspiratory Pressure (cm H2O) | over the first 5 minutes of life
Time to reach heart rate >100 beats per minute (seconds) | over the first 5 minutes of life
Time oxygen saturation within and outside of target range (seconds) | over the first 5 minutes of life
Time of the resuscitation (minutes) | up to 30 minutes of life
Time to demonstrate cycling of end tidal CO2 (seconds) | First minute of life
  Evaluated by analysis of video recording
Maximum End Tidal CO2 (mm Hg) | up to 30 minutes of life
Intubation (yes/no) in DR/NICU and age (hours) | up to 7 days of life
Surfactant (yes/no) in DR/NICU and age (hours) | up to 7 days of life
SVC Flow (ml/kg/min) | target time 6 hours of life
  plus/minus 6 hours
Right ventricular output (ml/kg/min) | 6 hours of life
  plus/minus 6 hours
Cardiac Output by Electrical Cardiometry (ml/kg/min) | over the first 24 hours of life
Cerebral StO2 by Near-Infrared Spectroscopy | over the first 24 hours of life
Fractional Oxygen Extraction by Near-Infrared Spectroscopy | 24 hours of life
Color Doppler diameter of ductus arteriosus shunt (mm) | 6 hours of life
  plus/minus 6 hours
Pulsed or continuous wave Doppler assessment of ductus arteriosus shunt direction (%time right to left) and velocity (m/s) | 6 hours of life
  plus/minus 6 hours
Color Doppler diameter of inter-atrial shunt (mm) | 6 hours of life
  plus/minus 6 hours
Pulsed and continuous wave Doppler assessment of inter-atrial shunt direction (% time right to left) and velocity (m/s) | 6 hours of life
  plus/minus 6 hours
Peak velocity of the tricuspid regurgitation jet (m/sec) (to calculate arterial pressure) | 6 hours of life
  plus/minus 6 hours
Record Blood pressure (SBP/DBP, MAP) and whether hypotensive (defined as < GA on DOL 1) yes/no | over the first 6 hours of life
Arterial and venous cord pH | at birth (first minute of life)
Peak total serum bilirubin (mg/dL) | participants will be followed for the duration of hospital stay, an expected average of 48 weeks
Duration of phototherapy days | participants will be followed for the duration of hospital stay, an expected average of 48 weeks
Serum hematocrit | at birth, 12 hours, and 30 days of life
Admission temperatures (degree Centigrade) | within 1 hour of life
Urine output (ml/kg/day) | over the first 72 hours
Mean Arterial Blood pressure (mm Hg) | over the first 24 hours
Use of cardiac inotropes (dopamine, dobutamine, epinephrine) (yes/no) hypotension | over the first 72 hours
Use of postnatal steroids (yes/no) | 4 months or until hospital discharge
Presence of intraventricular hemorrhage (yes/no) | participants will be followed for the duration of hospital stay, an expected average of 48 weeks
Presence of severe intraventricular hemorrhage (Grade 3 or 4) (yes/no) | 4 months or until hospital discharge
Presence of PVL (yes/no) | participants will be followed for the duration of hospital stay, an expected average of 48 weeks
Mortality (yes/no) | participants will be followed for the duration of hospital stay, an expected average of 48 weeks
Placental Weight | weighed within 24 hours of delivery of the infant
Maternal Hemoglobin | in the first 48 hours post delivery of the infant
Mean Airway Pressure (MAP) | First 5 minutes of life
Duration of CPAP or PPV | First one minute of life
  Evaluated by analysis of video recording
Length of umbilical cord allows use of LifeStart bed | First one minute of life
  Evaluated by analysis of video recording

CONTACTS AND LOCATIONS:
Overall Officials: Anup C Katheria, MD, Principal Investigator — Sharp HealthCare
Locations (1):
- Sharp Mary Birch Hospital for Women and Newborns, San Diego, California, United States

REFERENCES:
- [Derived] Katheria A, Poeltler D, Durham J, Steen J, Rich W, Arnell K, Maldonado M, Cousins L, Finer N. Neonatal Resuscitation with an Intact Cord: A Randomized Clinical Trial. J Pediatr. 2016 Nov;178:75-80.e3. doi: 10.1016/j.jpeds.2016.07.053. Epub 2016 Aug 26. PMID 27574999